CLINICAL TRIAL: NCT00837109
Title: Randomized Clinical Trial of Imagery Rescripting Treatment In Veterans With Trauma-Related Nightmares And Posttraumatic Stress Disorder (PTSD)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Primary investigator is no longer a part of the VA
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Long, Mary - Principal Investigator, Department of Veterans Affairs
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-24172
Record Dates: First submitted 2009-02-03; First posted 2009-02-05 (Estimated); Last update posted 2010-09-29 (Estimated); Status verified 2010-09

CONDITIONS: Stress Disorders, Post-Traumatic; Sleep Disorders
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Sleep Wake Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Imagery Rescripting Nightmare Treatment
  Interventions: Behavioral: Veteran Nightmare Treatment
- 2 (Active Comparator): Treatment-as-usual in the Trauma Recovery Program
  Interventions: Behavioral: Treatment-as-usual

INTERVENTIONS:
Behavioral: Veteran Nightmare Treatment — Veteran Nightmare Treatment Using Imagery Rescripting
  Arms: 1
Behavioral: Treatment-as-usual — Treatment-as-usual in the Trauma Recovery Program (that does not specifically target PTSD symptoms)
  Arms: 2

SUMMARY:
Research shows that symptoms of posttraumatic stress disorder (PTSD) are particularly high in veterans, and that trauma-related nightmares and sleep disturbances are common in veterans with PTSD. This is of concern because people with these problems will often use unhealthy ways of coping. Although trauma-related nightmares and difficulty sleeping are highly distressing, there are helpful treatments that do not involve taking medication. One of these treatments teaches specific skills to help people improve their sleep habits and to change their nightmares so that they are less upsetting. This treatment can be very helpful and research shows that people experience decreases in the frequency and severity of their nightmares, decreased symptoms of depression and PTSD, and improved sleep quality and quantity after completing treatment. However, because this treatment has only been studied with civilians, it is not clear how well this treatment works for veterans.

ELIGIBILITY:
Inclusion Criteria:

Participants will be:

1. patients at the VA in the Trauma Recovery Program;
2. English-speaking;
3. reporting at least one Posttraumatic Nightmare in the past week (due to any type of trauma);
4. have an existing PTSD International Classification of Diseases, Ninth Revision, Clinical Modification (ICD-9-CM); and
5. consenting to be randomized into treatment.

In addition, patients must agree to allow their assessment and therapy sessions to be video/audiotaped for the purposes of supervision and treatment integrity ratings. Participants receiving other forms of group or individual psychotherapy and/or psychotropic medication are eligible for the nightmare treatment condition of the study, provided that those interventions do not specifically target nightmares or PTSD. Thus, the study interventions will be in addition to standard care, except as indicated above.

Exclusion Criteria:

Patients

1. with current active suicidal/homicidal ideation and intent;
2. with current substance dependence;
3. a diagnosis of bipolar or psychosis; 4) prescribed the medication Prazosin (a psychotropic medication for the treatment of nightmares).

Patients in the nightmare treatment condition of the study will also be excluded if they are actively participating in another psychosocial treatment directly addressing their PTSD symptoms. Patients will not be excluded if they are taking psychotropic medication (except for Prazosin) and may continue to take their medication as prescribed throughout the study.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2009-02; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Posttraumatic Stress Symptom Scale-Self-Report (PSS-SR), Beck Depression Inventory-II (BDI-II) | Baseline, prior to each session, post-assessment, 3-month follow-up

SECONDARY OUTCOMES:
Posttraumatic Cognitions Inventory (PTCI) | Baseline, post-assessment, 3-month follow-up
Pittsburgh Sleep Quality Index-Addendum for PTSD (PSQI), | Baseline, post-assessment, 3-month follow-up
Trauma Related Nightmare Survey (TRNS) | Baseline, post-assessment, 3-month follow-up
Clinician-Administered PTSD Scale (CAPS) | Baseline, post-assessment, 3-month follow-up
Modules of the Mini-International Neuropsychiatric Interview (MINI) | Baseline
Treatment Evaluation Inventory (TEI) | Post-assessment
Client Satisfaction Questionnaire (CSQ) | Post-assessment

CONTACTS AND LOCATIONS:
Overall Officials: Mary E. Long, PhD, Principal Investigator — Michael E. DeBakey VA Medical Center (152)
Locations (1):
- Michael E. DeBakey VA Medical Center (152), Houston, Texas, United States